CLINICAL TRIAL: NCT05417126
Title: A Phase 2a, Open Label Multicenter Clinical Trial to Evaluate the Safety and Effects of a Single Intravitreal Injection of vMCO-010 Optogenetic Therapy in Subjects With Stargardt Disease
Brief Title: Safety and Effects of a Single Intravitreal Injection of vMCO-010 Optogenetic Therapy in Subjects With Stargardt Disease
Acronym: STARLIGHT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nanoscope Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTXMCO-004
Record Dates: First submitted 2022-06-09; First posted 2022-06-14 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Stargardt Disease
Keywords: Eye Diseases; Retinal Degeneration; Retinal Dystrophy; Eye Diseases, Hereditary
MeSH Terms: conditions — Stargardt Disease; Eye Diseases; Retinal Degeneration; Retinal Dystrophies; Eye Diseases, Hereditary

STUDY DESIGN:
Intervention Model Description: 6 subjects will be enrolled for vMCO-010 treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental-vMCO-010 (Experimental): Participants receive 1.2E11gc/eye of vMCO-010
  Interventions: Biological: Gene Therapy-vMCO-010

INTERVENTIONS:
Biological: Gene Therapy-vMCO-010 — The vMCO-010 is an adeno-associated virus serotype 2-based vector carried multi-characteristic opsin (MCO) gene expression cassette

SUMMARY:
The purpose of the study is to evaluate the safety and effects of a single intravitreal injection of virally-carried Multi-Characteristic Opsin (vMCO-010) in Subjects with Stargardt Disease

DETAILED DESCRIPTION:
This multicenter open label study will evaluate single dose level of vMCO-010 in up to 6 subjects with Stargardt's Disease. Subjects with documented clinical diagnosis of Stargardt disease (classic fleck phenotype and/or well-demarcated sub-foveal area of significantly reduced autofluorescence as imaged by FAF), or genetic diagnosis with pathogenic variants in ABCA4, ELOVL4, or PROM 1. All subjects will continue to be assessed for 48 weeks following treatment with vMCO-010.

ELIGIBILITY:
Inclusion Criteria:

1. ≥16 years of age
2. Able to comprehend and give informed consent.
3. Able to comply with testing and all protocol tests.
4. Documented clinical diagnosis of Stargardt disease (classic fleck phenotype and/or well-demarcated sub-foveal area of significantly reduced autofluorescence as imaged by FAF), or genetic diagnosis with pathogenic variants in ABCA4, ELOVL4, or PROM1
5. In the study eye: ETDRS BCVA in range of 1.3 logMAR (Approximate Snellen equivalent: 20/400) to 1.9 logMAR (Snellen equivalent: 20/1600), and ETDRS BCVA no better than 20/200 in the fellow eye.
6. Presence of retinal inner nuclear and nerve fiber layers on optical coherence tomography (OCT) testing in the study eye at screening

Exclusion Criteria:

1. Presence of any concurrent ocular disease that would affect study outcomes (e.g., severe cataracts; subjects can be enrolled 3 months after successful cataract surgery).
2. Received any of the following treatments: gene therapy, stem cell therapy, surgical implantation of prosthetic retinal chips (such as ARGUS-II) or sub-retinal injections.
3. Has taken non-approved items (supplement containing vitamin A or beta-carotene, liver-based products, or prescription oral retinoid medications) over the past 30 days
4. Participation in an interventional study of a vitamin A derivative ≤ 3 months prior to screening
5. Presence of significant cardiovascular or cerebrovascular disease, including stroke within 12 months of entry.
6. Resting heart rate outside specified limits upon repeated measurement.
7. History of uncontrolled diabetes, hepatitis, pancreatitis, cirrhosis, liver failure, uncontrolled thyroid disease or hypervitaminosis A.
8. Any intraocular surgery or thermal laser within 3 months of trial entry or any prior thermal laser in the macular region.
9. Any major surgical procedure within one month of trial entry or anticipated during the trial.
10. Clinically significant abnormal lab results at screening
11. Known serious allergies to the fluorescein dye used in angiography or intraocular pressure measurement, povidone iodine, or to the components of the vMCO-010 formulation
12. In the Investigator's opinion, any severe acute or chronic medical condition, psychiatric condition, physical examination finding or laboratory abnormality
13. Pre-existing conditions in the study eye such as glaucoma, diseases affecting the optic nerve causing significant visual field loss, history of uveitis, corneal or lenticular opacities).
14. Presence of any complicating systemic diseases such as malignancies whose treatment could affect central nervous system function..
15. Subjects who are positive for syphilis, hepatitis B, C, and human immunodeficiency virus (HIV) will be excluded..
16. Presence of narrow iridocorneal angles contraindicating pupillary dilation in the study eye.
17. Presence of disorders of the ocular media in the study eye which could interfere with visual acuity and other ocular assessments, including OCT, during the study period.
18. Presence of macular hole in the study eye, evident by ophthalmoscopy and/or by OCT examinations
19. Current evidence of retinal detachment in the study eye assessed by the Investigator that significantly affects central vision.
20. Current use of hydroxychloroquine, chloroquine, or any related retina-toxic compounds.
21. Active ocular inflammation or recurrent history of idiopathic or autoimmune associated uveitis.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Type, severity, and incidence of ocular and systemic adverse events (AEs) | 48 weeks
  Type, severity, and incidence of ocular and systemic adverse events (AEs), specifically those related to intravitreal injection of vMCO-010

SECONDARY OUTCOMES:
Effect of vMCO-010 as assessed by visual acuity | 48 weeks
  Change from baseline in BCVA at Weeks 12, 24, 48 in the study eye and the fellow eye
Effect of vMCO-010 on Light-guided Mobility | 48 Weeks
  Change from baseline in Multi-Luminance Mobility Test at weeks 12, 24, 48 in the study eye and the fellow eye
Effect of vMCO-010 on determination of shape | 48 Weeks
  Change from baseline in accuracy in determination of shape using Low Vision Multi-Parameter Test (LVMPT) at weeks 12, 24, 48 in the study eye and the fellow eye
Effect of vMCO-010 on determination of optical flow | 48 Weeks
  Change from baseline in accuracy in determination of optical flow using the LVMPT at weeks 12, 24 and 48 in the study eye and the fellow eye

CONTACTS AND LOCATIONS:
Overall Officials: Dr Samarendra Mohanty, Study Director — Nanoscope Therapeutics Inc.
Locations (2):
- United States (2):
  - Nanoscope Clinical Site, Miami, Florida
  - Nanoscope Clinical Site, McAllen, Texas

IPD SHARING:
Plan to Share IPD: Yes
The results of the clinical trial will be made available when the study is completed. The results will be published on this site and be available to conference presentations and publications.
Time Frame: Within 12 Months of study completion
Access Criteria: Safety and efficacy Results